CLINICAL TRIAL: NCT00001816
Title: The Impact of Starbright World on Children Being Treated at the NIH
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990105; 99-C-0105
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-05

CONDITIONS: Child, Hospitalized
Keywords: Anger; Loneliness; Mood; Psychosocial; Virtual Network

SUMMARY:
This study seeks to evaluate the impact of Starbright World (SBW) on hospitalized children. SBW is a virtual environment designed to link seriously ill children into an interactive online community where they can play games, learn about their condition, or talk with other ill children who are connected to the network. Our outcome evaluation of SBW will include assessments of pain, mood (anxious, depressed and energetic), anger, loneliness, and willingness to return to the NIH for treatment of children who are being treated at NIH. They will be assessed while engaging in "normal" recreational activities (in one of two available playrooms) and while using Starbright World. In addition, we will conduct a process evaluation of the implementation of Starbright World.

DETAILED DESCRIPTION:
This study seeks to evaluate the impact of Starbright World (SBW) on hospitalized children. SBW is a virtual environment designed to link seriously ill children into an interactive online community where they can play games, learn about their condition, or talk with other ill children who are connected to the network. Our outcome evaluation of SBW will include assessments of pain, mood (anxious, depressed and energetic), anger, loneliness, and willingness to return to the NIH for treatment of children who are being treated at the NIH. They will be assessed while engaging in "normal" recreational activities (in one of two available playrooms) and while using Starbright World. In addition, we will conduct a process evaluation of the implementation of Starbright World.

ELIGIBILITY:
Children between the ages of 8 and 21.

Currently on active protocol at NIH.

Access to playrooms on the 9th, 11th, 13th, and 14th floors.

Ability to read and understand English.

No presence of mental illness.

Ability to understand and/or perform tasks involved in using Starbright World.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35
Dates: Start 1999-05; Study Completion 2001-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bieri D, Reeve RA, Champion DG, Addicoat L, Ziegler JB. The Faces Pain Scale for the self-assessment of the severity of pain experienced by children: development, initial validation, and preliminary investigation for ratio scale properties. Pain. 1990 May;41(2):139-150. doi: 10.1016/0304-3959(90)90018-9. PMID 2367140
- [Background] Brennan PF, Moore SM, Smyth KA. The effects of a special computer network on caregivers of persons with Alzheimer's disease. Nurs Res. 1995 May-Jun;44(3):166-72. PMID 7761293
- [Background] Izenberg N, Lieberman DA. The Web, communication trends, and children's health. Part 4: How children use the Web. Clin Pediatr (Phila). 1998 Jun;37(6):335-40. doi: 10.1177/000992289803700601. PMID 9637896